CLINICAL TRIAL: NCT02252289
Title: Fluctuation of Airway Function in Children With Asthma Phenotype as a Predictor of Outcome
Brief Title: Fluctuation of Airway Function in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 154768; P2SKP3_151971/1 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Asthma; children; fluctuation analysis; exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Problematic severe asthmatics: Approximately 75 Children aged 5 to 17 years with problematic severe asthma (PSA). Two groups of PSA children will be recruited: those who have already been assessed as part of the Difficult Asthma protocol and classified as DA (difficult asthma)/ STRA (severe therapy resistant asthma) (training set) and those newly referred to the protocol (validation set).
  Previous enrolment or new referral to the Royal Brompton Hospital Difficult Asthma Protocol.
- Control group of moderate asthmatics: A control group of 30 children aged 5 to 17 years with mild to moderate asthma.

SUMMARY:
It is increasingly recognised that asthma is not a single disease but that there are many different phenotypes. Much of the work that we have previously carried out has focussed on differentiating children with difficult asthma (those whose asthma control improves with attention to the basics of asthma management such as adherence) from those with severe therapy resistant asthma (ongoing poor control despite high dose treatment and attention to the basics. Our collaborators in Basel, Switzerland have demonstrated that serial measurements of lung function (peak flow) in adults can characterise the severe asthma phenotype and its stability in adults with asthma. We plan to carry out twice daily peak flow measurement sin children with asthma using an electronic peak flow meter. We will analyse peak flow patterns in children with severe therapy resistant asthma (STRA), difficult asthma (DA) and mild to moderate asthma. We will also investigate the relationship between peak flow variations and symptoms, recorded in a daily diary and medication use, recorded by an electronic measuring device which attaches to the child's own inhaler (Smart-inhaler).

DETAILED DESCRIPTION:
Many children present with poorly controlled asthma despite high intensity treatment including high doses of inhaled steroids. A number of these children will get better once the basics of asthma management are addressed (such as adherence, allergen avoidance, smoking cessation). The remainder will need further escalation of treatment (with attendant side effects) and more invasive, investigations. Adults with severe asthma have been found to have differences in the fluctuation patterns of peak flow compared to mild asthmatics. This study will enable us to evaluate whether the same is true in children, enabling us to improve the way we identify children with difficult asthma (DA) and severe therapy resistant asthma (STRA) and whether the difficult asthma: DA group are in fact more similar to the mild/moderate group.

Asthma exacerbations are a serious and concerning problem in children with asthma. This study will enable us to assess whether mathematical modelling of fluctuation patterns can enable us to predict n asthma attack and therefore intervene before it becomes severe or even life threatening. This study will also enable us to investigate the relationship between symptoms, peak flow patterns, exacerbations and adherence to inhaled corticosteroids (ICS) as measured by electronic recording devices (Smart-inhalers).

This is an observational cohort study. If the child and their family are happy to participate in the study the first study visit can take place immediately. If they would like time to consider the study it can be deferred until their next routine attendance at the hospital.

Study visit 1:

Information will be collected relating to past medical history, asthma history and current medications (this information may also be obtained from the case notes).

The following standardised questionnaires will be used: Asthma Control Test, children >12 years (ACT) or Childhood Asthma Control Test, children 6-11years (cACT) (usually completed as part of a routine clinical visit); Mini Paediatric Asthma Quality of Life Questionnaire (PAQLQ); Medicines Adherence Rating Scale (MARS); Beliefs about Medicines Questionnaire (BMQ).

Study procedures:

Lung function (included as part of a routine clinic visit), bronchodilator reversibility (lung function repeated after administration of salbutamol), exhaled nitric oxide.

The child and their family will be issued with a paper diary, electronic peak flow meter (PIKO) and electronic monitoring device for their inhaler (Smart-inhaler) and shown how to use these.

Between visits:

Children will be asked to measure their peak flow twice daily (morning and evening) and record their symptoms in a diary. Their parents will also be asked to complete the diary. They will be contacted by the study investigator to check whether there are any technical problems and as a reminder to make the peak flow measurements and complete the diary.

Visit 2, approximately 12 weeks later (from 8 to 16 weeks)

The second study visit will be scheduled at the time of a planned hospital appointment. This will largely be a repeat of visit 1:

Information will be collected relating to asthma control and exacerbations since visit 1. The following standardised questionnaires will be used: Asthma Control Test, children >12 years (ACT) or Childhood Asthma Control Test, children 6-11years (cACT) (usually completed as part of a routine clinical visit); Mini Paediatric Asthma Quality of Life Questionnaire (PAQLQ)

Study procedures:

Lung function (included as part of a routine clinic visit), bronchodilator reversibility (lung function repeated after administration of salbutamol), exhaled nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* Parent / guardian must be able to give written informed consent prior to participation in the study, which includes ability to comply with the requirements and restrictions listed in the consent form. Informed consent must be obtained prior to undertaking any study procedures.
* Assent should be obtained from all children in the study where appropriate.
* Male or female subject aged between 5 - 17 years inclusive at screening.
* The parent / guardian, or where appropriate the child must be able to read, comprehend, and write at a sufficient level to complete study related materials.

Exclusion Criteria:

1. As a result of medical interview, physical examination or screening investigation the physician responsible considers the child unfit for the study.
2. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
3. Significant alternative diagnoses that may mimic or complicate asthma, in particular dysfunctional breathing, panic attacks, and overt psychosocial problems (if these are thought to be the major problem rather than in addition to severe asthma)
4. Significant other primary pulmonary disorders in particular cystic fibrosis, interstitial lung disease
5. Participants with bronchiectasis should only be excluded if this is thought to be the major pulmonary disorder rather than in addition to severe asthma

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with problematic severe asthma (PSA) will be identified from clinical records and the existing clinical database which records all those who have been assessed as part of the Difficult Asthma (DA) protocol. Children newly referred to the DA protocol will be identified by notification from Clinical Nurse Specialists (CNSs) who receive the referrals. Children with mild-moderate asthma will be identified from clinical records only.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Individual variability in peak expiratory flow | 3 months

SECONDARY OUTCOMES:
Individual variability in FEV1 | 3 months
Exacerbations (severe and moderate) | 3 months
Asthma control (asthma control test (ACT) scores ) | 3 months
ICS dose | 3 months
  Dose of inhaled corticosteroids
Asthma related quality of life (paediatric quality of life PAQLQ scores) | 3 months
Lung function (FEV1, bronchodilator reversibility) | 3 months
Adherence | 3 months
  Adherence as measured by Smart-inhaler data which will be downloaded at the follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Louise Fleming, MD, MBChB, Principal Investigator — Senior Lecturer Paediatric Respiratory Medicine, Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in children with asthma. Qual Life Res. 1996 Feb;5(1):35-46. doi: 10.1007/BF00435967. PMID 8901365
- [Background] Cohen JL, Mann DM, Wisnivesky JP, Home R, Leventhal H, Musumeci-Szabo TJ, Halm EA. Assessing the validity of self-reported medication adherence among inner-city asthmatic adults: the Medication Adherence Report Scale for Asthma. Ann Allergy Asthma Immunol. 2009 Oct;103(4):325-31. doi: 10.1016/s1081-1206(10)60532-7. PMID 19852197
- [Background] Menckeberg TT, Bouvy ML, Bracke M, Kaptein AA, Leufkens HG, Raaijmakers JA, Horne R. Beliefs about medicines predict refill adherence to inhaled corticosteroids. J Psychosom Res. 2008 Jan;64(1):47-54. doi: 10.1016/j.jpsychores.2007.07.016. PMID 18157999
- [Background] Frey U, Brodbeck T, Majumdar A, Taylor DR, Town GI, Silverman M, Suki B. Risk of severe asthma episodes predicted from fluctuation analysis of airway function. Nature. 2005 Dec 1;438(7068):667-70. doi: 10.1038/nature04176. PMID 16319891
- [Background] Bracken M, Fleming L, Hall P, Van Stiphout N, Bossley C, Biggart E, Wilson NM, Bush A. The importance of nurse-led home visits in the assessment of children with problematic asthma. Arch Dis Child. 2009 Oct;94(10):780-4. doi: 10.1136/adc.2008.152140. Epub 2009 Jun 21. PMID 19546102